CLINICAL TRIAL: NCT01794143
Title: Glycemia Reduction Approaches in Diabetes: A Comparative Effectiveness Study
Brief Title: A Comparative Effectiveness Study of Major Glycemia-lowering Medications for Treatment of Type 2 Diabetes
Acronym: GRADE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GRADE Study Group (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); National Heart, Lung, and Blood Institute (NHLBI) (NIH); Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GRADE; 1U01DK098246-01 (NIH)
Record Dates: First submitted 2013-02-13; First posted 2013-02-18 (Estimated); Results first posted 2026-02-10 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-01

CONDITIONS: Type 2 Diabetes; Comparative Effectiveness of Glycemia-lowering Medications
Keywords: Treatment of Type 2 diabetes; Comparative effectiveness research; Clinical trial; Patient-centered outcomes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Sulfonylurea Compounds; glimepiride; Dipeptidyl-Peptidase IV Inhibitors; Sitagliptin Phosphate; Liraglutide; Insulin Glargine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Sulfonylurea (glimepiride) (Active Comparator): Sulfonylurea
  Interventions: Drug: Sulfonylurea (glimepiride)
- DPP-4 inhibitor (Active Comparator): DPP-4 inhibitor (sitagliptin)
  Interventions: Drug: DPP-4 inhibitor (sitagliptin)
- GLP-1 receptor agonist (Active Comparator): GLP-1 receptor agonist (liraglutide)
  Interventions: Drug: GLP-1 receptor agonist (liraglutide)
- Insulin (glargine) (Active Comparator): Insulin (glargine), Lantus
  Interventions: Drug: Insulin (glargine)

INTERVENTIONS:
Drug: Sulfonylurea (glimepiride) — Used in accordance with labeling and/or usual practice.
  Other Names: Glimepiride
  Arms: Sulfonylurea (glimepiride)
Drug: DPP-4 inhibitor (sitagliptin) — Used in accordance with labeling and/or usual practice
  Other Names: Sitagliptin
  Arms: DPP-4 inhibitor
Drug: GLP-1 receptor agonist (liraglutide) — Used in accordance with labeling and/or usual practice.
  Other Names: Liraglutide
  Arms: GLP-1 receptor agonist
Drug: Insulin (glargine) — Used in accordance with labeling and/or usual practice.
  Other Names: Lantus
  Arms: Insulin (glargine)

SUMMARY:
The GRADE Study is a pragmatic, unmasked clinical trial that will compare commonly used diabetes medications, when combined with metformin, on glycemia-lowering effectiveness and patient-centered outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. Men or women diagnosed with diabetes at age ≥ 30 years (≥ 20 for American Indians)
2. Duration of diagnosed diabetes < 10 years
3. HbA1c criteria (at final run-in visit, ~2 weeks prior to randomization): 6.8-8.5%
4. Taking a daily dose of ≥ 1000 mg metformin for a minimum of 8 weeks at final run-in
5. Willingness to administer daily subcutaneous injections, take a second diabetes drug after randomization, potentially initiate insulin and intensify insulin therapy if study metabolic goals are not met, perform self-monitoring of blood glucose
6. Fluent in either English or Spanish
7. A negative pregnancy test for all females of childbearing potential (i.e. pre-menopausal, and not surgically sterile)
8. Provision of signed and dated informed consent prior to any study procedures

Exclusion Criteria:

1. Suspected type 1 diabetes (lean with polyuria, polydipsia, and weight loss with little response to metformin) or "secondary" diabetes due to specific causes (e.g. previously diagnosed monogenic syndromes, pancreatic surgery, pancreatitis)
2. Current or previous (within past 6 months) treatment with any diabetes drug/glucose-lowering medication other than metformin (limited use of no longer than seven days is allowed, for example during hospitalization)
3. More than 10 years of treatment with metformin at time of randomization screening
4. History of intolerance or allergy or other contraindications to any of the proposed study medications
5. Resides in the same household with another GRADE study participant
6. Current need for any specific glucose-lowering medications solely for other conditions, for example for polycystic ovary syndrome
7. Symptomatic hyperglycemia requiring immediate therapy during screening or run-in, in the judgment of the physician
8. A life-threatening event within 30 days prior to screening or currently planned major surgery
9. Any major cardiovascular event in previous year, including history of myocardial infarction, stroke, or vascular procedure such as coronary artery or peripheral bypass grafting, stent placements (peripheral or coronary) or angioplasty.
10. Plans for pregnancy during the course of the study for women of child-bearing potential
11. History of or planning bariatric surgery, including banding procedures or surgical gastric and/or intestinal bypass (if banding removed, may be considered eligible after 1 year)
12. History of congestive heart failure (NYHA 3 or greater)
13. History of pancreatitis
14. History of cancer, other than non-melanoma skin cancer, that required therapy in the 5 years prior to randomization
15. Personal or family history of MEN-2 or family history of medullary thyroid cancer
16. Estimated GFR (eGFR) <30 ml/min/1.73 m2 or end stage renal disease requiring renal replacement therapy
17. History of severe liver disease or acute hepatitis or ALT > 3 times upper limit of normal
18. Current alcoholism or excessive alcohol intake
19. Previous organ transplant
20. Treatment with oral or systemic glucocorticoids (other than short-term treatment, for example for poison ivy) or disease likely to require periodic or regular glucocorticoid therapy (inhaled steroids are allowed)
21. Treatment with atypical antipsychotics
22. History of hemolytic anemia, chronic transfusion requirement, or other condition rendering HbA1c results unreliable as indicator of chronic glucose levels, or hematocrit <35 for males and <33 for females
23. Clinically or medically unstable with expected survival <1 year
24. Unwillingness to permit sites to contact the PCP to communicate information about the study and the participant's data
25. No non-study PCP or inability to identify such a PCP (who will provide non-study care) by the time of final run-in
26. Participation in another interventional clinical trial
27. Previous randomization in the GRADE study
28. In the opinion of the principal investigator (PI), any other factor, including language barrier, likely to limit compliance with the protocol

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7850 (Actual)
Dates: Start 2013-05; Primary Completion 2021-04-30 (Actual); Study Completion 2021-04-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David M Nathan, MD, Study Chair — Massachusetts General Hospital
Locations (36):
- United States (36):
  - University of Alabama-Birmingham, Birmingham, Alabama
  - Southwestern American Indian Center, Phoenix, Arizona
  - Veterans Medical Research Foundation, San Diego (San Diego VA), San Diego, California
  - University of Colorado, Denver, Colorado
  - Yale University School of Medicine, New Haven, Connecticut
  - South Florida VA Foundation (Miami VA), Miami, Florida
  - Atlanta VA Medical Center, Decatur, Georgia
  - Kaiser Permanente of Georgia, Duluth, Georgia
  - Pacific Health Research and Education Institute (VA Pacific Islands), Honolulu, Hawaii
  - Indiana University School of Medicine, Indianapolis, Indiana
  - University of Iowa, Iowa City, Iowa
  - Pennington Biomedical Research Center, Baton Rouge, Louisiana
  - MedStar Health Research Institute, Hyattsville, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - International Diabetes Center, Minneapolis, Minnesota
  - University of Minnesota, Minneapolis, Minnesota
  - Washington University School of Medicine, St Louis, Missouri
  - University of Nebraska, Omaha, Nebraska
  - University of New Mexico School of Medicine, Albuquerque, New Mexico
  - State University of New York (SUNY)-Downstate Medical Center, Brooklyn, New York
  - Columbia University Naomi Berrie Diabetes Center, New York, New York
  - Mount Sinai St. Luke's Hospital, New York, New York
  - Albert Einstein College of Medicine, The Bronx, New York
  - Duke University Medical Center, Durham, North Carolina
  - University of North Carolina Diabetes Care Center, Durham, North Carolina
  - University of Cincinnati, Cincinnati, Ohio
  - Case Western Reserve University School of Medicine, Cleveland, Ohio
  - Kaiser Permanente Northwest, Portland, Oregon
  - Oregon Health and Science University, Portland, Oregon
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Baylor Endocrine Center, Dallas, Texas
  - University of Texas-Southwestern Medical Center, Dallas, Texas
  - Baylor College of Medicine, Houston, Texas
  - University of Texas Health Science Center, San Antonio, Texas
  - Seattle Institute for Biomedical and Clinical Research, Seattle, Washington

REFERENCES:
- [Background] Butera NM, Zeng D, Heiss G, Cai J. Modeling longitudinal change in biomarkers using data from a complex survey sampling design: An application to the Hispanic Community Health Study/Study of Latinos. Stat Med. 2023 Feb 28;42(5):632-655. doi: 10.1002/sim.9635. Epub 2023 Jan 11. PMID 36631123
- [Background] Butera NM, Zeng D, Green Howard A, Gordon-Larsen P, Cai J. A doubly robust method to handle missing multilevel outcome data with application to the China Health and Nutrition Survey. Stat Med. 2022 Feb 20;41(4):769-785. doi: 10.1002/sim.9260. Epub 2021 Nov 16. PMID 34786739
- [Background] Ghosh A, Chan W, Younes N, Davis BR. A Dynamic Risk Model for Multitype Recurrent Events. Am J Epidemiol. 2023 Apr 6;192(4):621-631. doi: 10.1093/aje/kwac213. PMID 36549905
- [Background] Lachin JM, Bebu I. Closed testing of each group versus the others combined in a multiple group analysis. Clin Trials. 2020 Feb;17(1):77-86. doi: 10.1177/1740774519879932. Epub 2019 Oct 24. PMID 31647326
- [Background] Bebu I, Lachin JM. Properties of composite time to first event versus joint marginal analyses of multiple outcomes. Stat Med. 2018 Nov 30;37(27):3918-3930. doi: 10.1002/sim.7849. Epub 2018 Jun 28. PMID 29956365
- [Background] Lachin JM, Bebu I. Application of the Wei-Lachin multivariate one-directional test to multiple event-time outcomes. Clin Trials. 2015 Dec;12(6):627-33. doi: 10.1177/1740774515601027. Epub 2015 Sep 2. PMID 26336199
- [Background] Lachin JM. Applications of the Wei-Lachin multivariate one-sided test for multiple outcomes on possibly different scales. PLoS One. 2014 Oct 17;9(10):e108784. doi: 10.1371/journal.pone.0108784. eCollection 2014. PMID 25329662
- [Background] Lachin JM. Fallacies of last observation carried forward analyses. Clin Trials. 2016 Apr;13(2):161-8. doi: 10.1177/1740774515602688. Epub 2015 Sep 22. PMID 26400875
- [Result] Pop-Busui R, Rosin SP, Butera NM, Krause-Steinrauf H, Abou Assi H, Garg RK, Inzucchi SE, Katona A, McGill JB, Mudaliar S, Schade DS, Seaquist ER, Tiktin M, Soliman EZ, Green JB; GRADE Research Group. Differences in Prevalence and Incidence of Electrocardiogram Abnormalities and Cardiovascular Autonomic Neuropathy Among Randomized Glucose-Lowering Treatments in Early Type 2 Diabetes: The Glycemia Reduction Approaches in Diabetes (GRADE) Cohort. Diabetes Care. 2025 Nov 1;48(11):1960-1970. doi: 10.2337/dc25-1087. PMID 40986645
- [Result] Presley CA, Butera NM, Krause-Steinrauf H, Desouza CV, Hollander PA, Hoogendoorn CJ, Lagari VS, Legowski EA, Martin CL, Rasouli N, Gonzalez JS, Cherrington AL. Lack of Association of Emotional Distress With Insulin Initiation in the GRADE Randomized Diabetes Comparative Effectiveness Trial. Sci Diabetes Self Manag Care. 2025 Aug;51(4):382-393. doi: 10.1177/26350106251361363. Epub 2025 Aug 1. PMID 40751289
- [Result] Hsia DS, Younes N, Ghosh A, Kazemi EJ, Krause-Steinrauf H, Buse JB, Baker C, Brown-Friday J, Diaz E, Diner J, Groessl EJ, Legowski EA, Mariash CN, Waltje AH, Wexler DJ, Martin CL; GRADE Research Group. Association of Hospitalizations With Randomized Glycemia-Lowering Treatment in GRADE. Diabetes Care. 2025 Jul 1;48(7):1288-1294. doi: 10.2337/dc24-2839. PMID 40424051
- [Result] Luchsinger JA, Rosin SP, Kazemi EJ, Younes N, Suratt CE, Fattaleh BN, Florez HJ, Gonzalez JS, Hollander P, Hox SH, Kuo S, Lee MS, Martens T, Pop-Busui R, Seaquist ER, Waltje AH, Barzilay JI; GRADE Research Group. Glucose-Lowering Medications, Glycemia, and Cognitive Outcomes: The GRADE Randomized Clinical Trial. JAMA Intern Med. 2025 Jul 1;185(7):778-787. doi: 10.1001/jamainternmed.2025.1189. PMID 40388190
- [Result] Wexler DJ, Garvey WT, Ghosh A, Kazemi EJ, Krause-Steinrauf H, Ahmann AJ, Brown-Friday J, Casula S, Cherrington AL, Elasy TA, Fortmann SP, Krakoff JA, Mudaliar S, Tiktin M, Younes N; GRADE Study Research Group. Weight Gain Was Associated With Worsening Glycemia and Cardiovascular and Kidney Outcomes in Patients With Type 2 Diabetes Independent of Diabetes Medication in the GRADE Randomized Controlled Trial. Diabetes Care. 2025 Jun 1;48(6):935-944. doi: 10.2337/dc24-2825. PMID 40267365
- [Result] Utzschneider KM, Tripputi M, Butera NM, Mari A, Rosin SP, Banerji MA, Bergenstal RM, Brown N, Carlson AL, DeFronzo RA, Gramzinski MR, Harindhanavudhi T, Kozedub A, Sivitz WI, Steffes MW, Balasubramanyam A, Rasouli N; GRADE Research Group. Differential Treatment Effects on beta-Cell Function Using Model-Based Parameters in Type 2 Diabetes: Results From the Glycemia Reduction Approaches in Diabetes: A Comparative Effectiveness Study (GRADE). Diabetes Care. 2025 Apr 1;48(4):623-631. doi: 10.2337/dc24-2419. PMID 39998948
- [Result] Nathan DM. Response to Comment on Nathan et al. Relationship Between Average Glucose Levels and HbA1c Differs Across Racial Groups: A Substudy of the GRADE Randomized Trial. Diabetes Care 2024;47:2155-2163. Diabetes Care. 2025 Mar 1;48(3):e34-e35. doi: 10.2337/dci24-0095. No abstract available. PMID 39977640
- [Result] Ehrmann D, Krause-Steinrauf H, Uschner D, Wen H, Hoogendoorn CJ, Crespo-Ramos G, Presley C, Arends VL, Cohen RM, Garvey WT, Martens T, Willis HJ, Cherrington A, Gonzalez JS; GRADE Research Group. Differential associations of somatic and cognitive-affective symptoms of depression with inflammation and insulin resistance: cross-sectional and longitudinal results from the Emotional Distress Sub-Study of the GRADE study. Diabetologia. 2025 Jul;68(7):1403-1415. doi: 10.1007/s00125-025-06369-8. Epub 2025 Feb 14. PMID 39951058
- [Result] Seaquist ER, Phillips LS, Ghosh A, Baker C, Bergenstal RM, Crandall JP, Goland RS, Gramzinski MR, Hox SH, Hsia DS, Johnson ML, Lachin JM, Raskin P, Valencia WM, Waltje AH, Younes N; GRADE Research Group. Glycemia reduction in type 2 diabetes-Hypoglycemia outcomes: A randomized clinical trial. PLoS One. 2024 Nov 15;19(11):e0309907. doi: 10.1371/journal.pone.0309907. eCollection 2024. PMID 39546502
- [Result] Nathan DM, Herman WH, Larkin ME, Krause-Steinrauf H, Abou Assi H, Ahmann AJ, Brown-Friday J, Hsia DS, Harindhanavudhi T, Johnson M, Arends VL, Butera NM, Rosin SP, Lachin JM, Younes N; GRADE Study Research Group. Relationship Between Average Glucose Levels and HbA1c Differs Across Racial Groups: A Substudy of the GRADE Randomized Trial. Diabetes Care. 2024 Dec 1;47(12):2155-2163. doi: 10.2337/dc24-1362. PMID 39312277
- [Result] Gonzalez JS, Bebu I, Krause-Steinrauf H, Hoogendoorn CJ, Crespo-Ramos G, Presley C, Naik AD, Kuo S, Johnson ML, Wexler D, Crandall JP, Bantle AE, Arends V, Cherrington AL; GRADE Research Group. Differential Effects of Type 2 Diabetes Treatment Regimens on Diabetes Distress and Depressive Symptoms in the Glycemia Reduction Approaches in Diabetes: A Comparative Effectiveness Study (GRADE). Diabetes Care. 2024 Apr 1;47(4):610-619. doi: 10.2337/dc23-2459. PMID 38416773
- [Result] Green JB, Everett BM, Ghosh A, Younes N, Krause-Steinrauf H, Barzilay J, Desouza C, Inzucchi SE, Pokharel Y, Schade D, Scrymgeour A, Tan MH, Utzschneider KM, Mudaliar S; GRADE Study Research Group. Cardiovascular Outcomes in GRADE (Glycemia Reduction Approaches in Type 2 Diabetes: A Comparative Effectiveness Study). Circulation. 2024 Mar 26;149(13):993-1003. doi: 10.1161/CIRCULATIONAHA.123.066604. Epub 2024 Feb 12. PMID 38344820
- [Result] Hampe CS, Shojaie A, Brooks-Worrell B, Dibay S, Utzschneider K, Kahn SE, Larkin ME, Johnson ML, Younes N, Rasouli N, Desouza C, Cohen RM, Park JY, Florez HJ, Valencia WM, Stempel R, Palmer JP, Balasubramanyam A. GAD65Abs Are Not Associated With Beta-Cell Dysfunction in Patients With T2D in the GRADE Study. J Endocr Soc. 2024 Feb 8;8(3):bvad179. doi: 10.1210/jendso/bvad179. eCollection 2024 Jan 16. PMID 38333889
- [Result] Hsia DS, Younes N, Krause-Steinrauf H, Kassem LS; GRADE Research Group. The incidence of retinopathy in the Glycemia Reduction Approaches in Diabetes: A Comparative Effectiveness study (GRADE). J Diabetes Complications. 2024 Mar;38(3):108692. doi: 10.1016/j.jdiacomp.2024.108692. Epub 2024 Feb 5. PMID 38354481
- [Result] Garvey WT, Cohen RM, Butera NM, Kazemi EJ, Younes N, Rosin SP, Suratt CE, Ahmann A, Hollander PA, Krakoff J, Martin CL, Seaquist E, Steffes MW, Lachin JM; GRADE Research Group. Association of Baseline Factors With Glycemic Outcomes in GRADE: A Comparative Effectiveness Randomized Clinical Trial. Diabetes Care. 2024 Apr 1;47(4):562-570. doi: 10.2337/dc23-1782. PMID 38285957
- [Result] Banerji MA, Buse JB, Younes N, Krause-Steinrauf H, Ghazi A, Lee M, Park J, Pop-Busui R, Underkofler C, Fortmann SP; GRADE Research Group. Mortality in the Glycemia Reduction Approaches in Diabetes: A Comparative Effectiveness Study (GRADE). Diabetes Care. 2024 Apr 1;47(4):589-593. doi: 10.2337/dc23-1356. PMID 38252886
- [Result] Cherrington AL, Bebu I, Krause-Steinrauf H, Hoogendoorn CJ, Crespo-Ramos G, Presley C, Naik AD, Balasubramanyam A, Gramzinski MR, Killean T, Arends VL, Gonzalez JS; GRADE Research Group. Does Emotional Distress Predict Worse Glycemic Control Over Time? Results From the Glycemia Reduction Approaches in Diabetes: A Comparative Effectiveness Study (GRADE). Diabetes Care. 2024 Apr 1;47(4):620-628. doi: 10.2337/dc23-0642. PMID 38252848
- [Result] Hoogendoorn CJ, Krause-Steinrauf H, Uschner D, Wen H, Presley CA, Legowski EA, Naik AD, Golden SH, Arends VL, Brown-Friday J, Krakoff JA, Suratt CE, Waltje AH, Cherrington AL, Gonzalez JS; GRADE Research Group. Emotional Distress Predicts Reduced Type 2 Diabetes Treatment Adherence in the Glycemia Reduction Approaches in Diabetes: A Comparative Effectiveness Study (GRADE). Diabetes Care. 2024 Apr 1;47(4):629-637. doi: 10.2337/dc23-1401. PMID 38227900
- [Result] Rasouli N, Younes N, Ghosh A, Albu J, Cohen RM, DeFronzo RA, Diaz E, Sayyed Kassem L, Luchsinger JA, McGill JB, Sivitz WI, Tamborlane WV, Utzschneider KM, Kahn SE; GRADE Research Group. Longitudinal Effects of Glucose-Lowering Medications on beta-Cell Responses and Insulin Sensitivity in Type 2 Diabetes: The GRADE Randomized Clinical Trial. Diabetes Care. 2024 Apr 1;47(4):580-588. doi: 10.2337/dc23-1070. PMID 38211595
- [Result] Kirkman MS, Tripputi M, Krause-Steinrauf H, Bebu I, AbouAssi H, Burch H, Duran-Valdez E, Florez H, Garvey WT, Hsia DS, Salam M, Pop-Busui R; GRADE Research Group. Comparative Effects of Randomized Second-line Therapy for Type 2 Diabetes on a Composite Outcome Incorporating Glycemic Control, Body Weight, and Hypoglycemia: An Analysis of the Glycemia Reduction Approaches in Diabetes: A Comparative Effectiveness Study (GRADE). Diabetes Care. 2024 Apr 1;47(4):594-602. doi: 10.2337/dc23-1332. PMID 38194519
- [Result] Utzschneider KM, Younes N, Butera NM, Balasubramanyam A, Bergenstal RM, Barzilay J, DeSouza C, DeFronzo RA, Elasy T, Krakoff J, Kahn SE, Rasouli N, Valencia WM, Sivitz WI; GRADE Research Group. Impact of Insulin Sensitivity and beta-Cell Function Over Time on Glycemic Outcomes in the Glycemia Reduction Approaches in Diabetes: A Comparative Effectiveness Study (GRADE): Differential Treatment Effects of Dual Therapy. Diabetes Care. 2024 Apr 1;47(4):571-579. doi: 10.2337/dc23-1059. PMID 38190619
- [Result] Cherrington AL, Tripputi MT, Younes N, Herman WH, Katona A, Groessl EJ, Craig J, Gonzalez JS, Garg R, Casula S, Kuo S, Florez HJ; GRADE Research Group. Impact of Glucose-Lowering Medications on Health-Related Quality of Life in the Glycemia Reduction Approaches in Diabetes: A Comparative Effectiveness Study (GRADE). Diabetes Care. 2024 Apr 1;47(4):603-609. doi: 10.2337/dc23-1648. PMID 38190625
- [Result] Hollander PA, Krause-Steinrauf H, Butera NM, Kazemi EJ, Ahmann AJ, Fattaleh BN, Johnson ML, Killean T, Lagari VS, Larkin ME, Legowski EA, Rasouli N, Willis HJ, Martin CL; GRADE Research Group. The Use of Rescue Insulin in the Glycemia Reduction Approaches in Diabetes: A Comparative Effectiveness Study (GRADE). Diabetes Care. 2024 Apr 1;47(4):638-645. doi: 10.2337/dc23-0516. PMID 37756542
- [Result] Crespo-Ramos G, Bebu I, Krause-Steinrauf H, Hoogendoorn CJ, Fang R, Ehrmann D, Presley C, Naik AD, Katona A, Walker EA, Cherrington A, Gonzalez JS; GRADE Research Group. Emotional distress and cardiovascular disease risk among participants enrolled in the Glycemia Reduction Approaches in Diabetes: A Comparative Effectiveness (GRADE) study. Diabetes Res Clin Pract. 2023 Sep;203:110808. doi: 10.1016/j.diabres.2023.110808. Epub 2023 Jun 30. PMID 37394014
- [Result] Luchsinger JA, Kazemi EJ, Sanchez DL, Larkin ME, Valencia WM, Desouza C, Carlson AL, Pop-Busui R, Seaquist ER, Florez HJ, Barzilay J; GRADE Research Group. BMI, insulin sensitivity, and cognition in early type 2 diabetes: The Glycemia Reduction Approaches in Diabetes: A Comparative Effectiveness Study. Obesity (Silver Spring). 2023 Jul;31(7):1812-1824. doi: 10.1002/oby.23785. PMID 37368512
- [Result] Cherrington AL, Krause-Steinrauf H, Aroda V, Buse JB, Fattaleh B, Fortmann SP, Hall S, Hox SH, Kuhn A, Killean T, Loveland A, Phillips LS, Jackson AU, Waltje A, McKee MD; GRADE Research Group. Use of comprehensive recruitment strategies in the glycemia reduction approaches in diabetes: A comparative effectiveness study (GRADE) multi-center clinical trial. Clin Trials. 2023 Oct;20(5):546-558. doi: 10.1177/17407745231175919. Epub 2023 Jun 17. PMID 37329282
- [Result] Wexler DJ, de Boer IH, Ghosh A, Younes N, Bebu I, Inzucchi SE, McGill JB, Mudaliar S, Schade D, Steffes MW, Tamborlane WV, Tan MH, Ismail-Beigi F; GRADE Research Group. Comparative Effects of Glucose-Lowering Medications on Kidney Outcomes in Type 2 Diabetes: The GRADE Randomized Clinical Trial. JAMA Intern Med. 2023 Jul 1;183(7):705-714. doi: 10.1001/jamainternmed.2023.1487. PMID 37213109
- [Result] Gulanski BI, Butera NM, Krause-Steinrauf H, Lichtman JH, Harindhanavudhi T, Green JB, Suratt CE, AbouAssi H, Desouza C, Ahmann AJ, Wexler DJ, Aroda VR; GRADE Research Group. Higher burden of cardiometabolic and socioeconomic risk factors in women with type 2 diabetes: an analysis of the Glycemic Reduction Approaches in Diabetes (GRADE) baseline cohort. BMJ Open Diabetes Res Care. 2023 Apr;11(2):e003159. doi: 10.1136/bmjdrc-2022-003159. PMID 37094945
- [Result] Seegmiller JC, Schmit DJ, Arends VL, Steffes MW, Kahn SE, Younes N; GRADE Research Group. Assessment of circulating insulin using liquid chromatography-mass spectrometry during insulin glargine treatment in type 2 diabetes: Implications for estimating insulin sensitivity and beta-cell function. Diabetes Obes Metab. 2023 Jul;25(7):1995-2004. doi: 10.1111/dom.15072. Epub 2023 Apr 24. PMID 36999229
- [Result] Gonzalez JS, Krause-Steinrauf H, Bebu I, Crespo-Ramos G, Hoogendoorn CJ, Naik AD, Waltje A, Walker E, Ehrmann D, Brown-Friday J, Cherrington A; GRADE Research Group. Emotional distress, self-management, and glycemic control among participants enrolled in the glycemia reduction approaches in diabetes: A comparative effectiveness (GRADE) study. Diabetes Res Clin Pract. 2023 Feb;196:110229. doi: 10.1016/j.diabres.2022.110229. Epub 2022 Dec 20. PMID 36549506
- [Result] GRADE Study Research Group; Nathan DM, Lachin JM, Bebu I, Burch HB, Buse JB, Cherrington AL, Fortmann SP, Green JB, Kahn SE, Kirkman MS, Krause-Steinrauf H, Larkin ME, Phillips LS, Pop-Busui R, Steffes M, Tiktin M, Tripputi M, Wexler DJ, Younes N. Glycemia Reduction in Type 2 Diabetes - Microvascular and Cardiovascular Outcomes. N Engl J Med. 2022 Sep 22;387(12):1075-1088. doi: 10.1056/NEJMoa2200436. PMID 36129997
- [Result] GRADE Study Research Group; Nathan DM, Lachin JM, Balasubramanyam A, Burch HB, Buse JB, Butera NM, Cohen RM, Crandall JP, Kahn SE, Krause-Steinrauf H, Larkin ME, Rasouli N, Tiktin M, Wexler DJ, Younes N. Glycemia Reduction in Type 2 Diabetes - Glycemic Outcomes. N Engl J Med. 2022 Sep 22;387(12):1063-1074. doi: 10.1056/NEJMoa2200433. PMID 36129996
- [Result] Aroda VR, Krause-Steinrauf K, Kazemi EJ, Buse JB, Gulanski BI, Florez HJ, Ahmann AJ, Loveland A, Kuhn A, Lonier JY, Wexler DJ, and the GRADE Research Group. Clinical and Metabolic Characterization of Adults With Type 2 Diabetes by Age in the Glycemia Reduction Approaches in Diabetes: A Comparative Effectiveness Study (GRADE) Cohort. Diabetes Care. July 13, 2022; doi: https://doi.org/10.2337/dc21-2659. PubMed Central PMID/PMCID: PMC9375440
- [Result] Florez HJ, Ghosh A, Pop-Busui R, Hox SH, Underkofler C, McKee MD, Park J, Rhee MK, Killean T, Krause-Steinrauf H, Aroda VR, Wexler DJ; GRADE Research Group. Differences in complications, cardiovascular risk factor, and diabetes management among participants enrolled at veterans affairs (VA) and non-VA medical centers in the glycemia reduction approaches in diabetes: A comparative effectiveness study (GRADE). Diabetes Res Clin Pract. 2022 Feb;184:109188. doi: 10.1016/j.diabres.2021.109188. Epub 2021 Dec 28. PMID 34971663
- [Result] Brooks-Worrell B, Hampe CS, Hattery EG, Palomino B, Zangeneh SZ, Utzschneider K, Kahn SE, Larkin ME, Johnson ML, Mather KJ, Younes N, Rasouli N, Desouza C, Cohen RM, Park JY, Florez HJ, Valencia WM; GRADE Beta-cell Ancillary Study Network; Shojaie A, Palmer JP, Balasubramanyam A. Islet Autoimmunity is Highly Prevalent and Associated With Diminished beta-Cell Function in Patients With Type 2 Diabetes in the Grade Study. Diabetes. 2022 Jan 21;71(6):1261-71. doi: 10.2337/db21-0590. Online ahead of print. PMID 35061024
- [Result] Nathan DM, Krause-Steinrauf H, Braffett BH, Arends VL, Younes N, McGee P, Lund C, Johnson M, Lorenzi G, Gao X, Steffes MW, Lachin JM; GRADE Research Group; DCCT/EDIC Research Group. Comparison of central laboratory HbA1c measurements obtained from a capillary collection versus a standard venous whole blood collection in the GRADE and EDIC studies. PLoS One. 2021 Nov 15;16(11):e0257154. doi: 10.1371/journal.pone.0257154. eCollection 2021. PMID 34780485
- [Result] Luchsinger JA, Younes N, Manly JJ, Barzilay J, Valencia W, Larkin ME, Falck-Ytter C, Krause-Steinrauf H, Pop-Busui R, Florez H, Seaquist E; GRADE Research Group; GRADE Research Group Investigators:. Association of Glycemia, Lipids, and Blood Pressure With Cognitive Performance in People With Type 2 Diabetes in the Glycemia Reduction Approaches in Diabetes: A Comparative Effectiveness Study (GRADE). Diabetes Care. 2021 Oct;44(10):2286-2292. doi: 10.2337/dc20-2858. Epub 2021 Jul 20. PMID 34285097
- [Result] Barzilay JI, Ghosh A, Busui RP, Ahmann A, Balasubramanyam A, Banerji MA, Cohen RM, Green J, Ismail-Beigi F, Martin CL, Seaquist E, Luchsinger JA; GRADE Research Group. The cross-sectional association of cognition with diabetic peripheral and autonomic neuropathy-The GRADE study. J Diabetes Complications. 2021 Dec;35(12):108047. doi: 10.1016/j.jdiacomp.2021.108047. Epub 2021 Sep 15. PMID 34556408
- [Result] Cherrington AL, Krause-Steinrauf H, Bebu I, Naik AD, Walker E, Golden SH, Gonzalez JS; GRADE Research Group. Study of emotional distress in a comparative effectiveness trial of diabetes treatments: Rationale and design. Contemp Clin Trials. 2021 Aug;107:106366. doi: 10.1016/j.cct.2021.106366. Epub 2021 Mar 22. PMID 33766761
- [Result] Utzschneider KM, Younes N, Rasouli N, Barzilay JI, Banerji MA, Cohen RM, Gonzalez EV, Ismail-Beigi F, Mather KJ, Raskin P, Wexler DJ, Lachin JM, Kahn SE; GRADE Research Group. Shape of the OGTT glucose response curve: relationship with beta-cell function and differences by sex, race, and BMI in adults with early type 2 diabetes treated with metformin. BMJ Open Diabetes Res Care. 2021 Sep;9(1):e002264. doi: 10.1136/bmjdrc-2021-002264. PMID 34531242
- [Result] Utzschneider KM, Younes N, Rasouli N, Barzilay J, Banerji MA, Cohen RM, Gonzalez EV, Mather KJ, Ismail-Beigi F, Raskin P, Wexler DJ, Lachin JM, Kahn SE; GRADE Research Group. Association of glycemia with insulin sensitivity and beta-cell function in adults with early type 2 diabetes on metformin alone. J Diabetes Complications. 2021 May;35(5):107912. doi: 10.1016/j.jdiacomp.2021.107912. Epub 2021 Mar 17. PMID 33752962
- [Result] Barzilay JI, Younes N, Pop-Busui R, Florez H, Seaquist E, Falck-Ytter C, Luchsinger JA; GRADE Research Group. The cross-sectional association of renal dysfunction with tests of cognition in middle-aged adults with early type 2 diabetes: The GRADE Study. J Diabetes Complications. 2021 Mar;35(3):107805. doi: 10.1016/j.jdiacomp.2020.107805. Epub 2020 Nov 26. PMID 33288412
- [Result] Rasouli N, Younes N, Utzschneider KM, Inzucchi SE, Balasubramanyam A, Cherrington AL, Ismail-Beigi F, Cohen RM, Olson DE, DeFronzo RA, Herman WH, Lachin JM, Kahn SE; GRADE Research Group. Association of Baseline Characteristics With Insulin Sensitivity and beta-Cell Function in the Glycemia Reduction Approaches in Diabetes: A Comparative Effectiveness (GRADE) Study Cohort. Diabetes Care. 2021 Feb;44(2):340-349. doi: 10.2337/dc20-1787. Epub 2020 Dec 17. PMID 33334808
- [Result] Mather KJ, Bebu I, Baker C, Cohen RM, Crandall JP, DeSouza C, Green JB, Kirkman MS, Krause-Steinrauf H, Larkin M, Pettus J, Seaquist ER, Soliman EZ, Schroeder EB, Wexler DJ, Pop-Busui R; GRADE Research Group. Prevalence of microvascular and macrovascular disease in the Glycemia Reduction Approaches in Diabetes - A Comparative Effectiveness (GRADE) Study cohort. Diabetes Res Clin Pract. 2020 Jul;165:108235. doi: 10.1016/j.diabres.2020.108235. Epub 2020 May 23. PMID 32450102
- [Result] Sivitz WI, Phillips LS, Wexler DJ, Fortmann SP, Camp AW, Tiktin M, Perez M, Craig J, Hollander PA, Cherrington A, Aroda VR, Tan MH, Krakoff J, Rasouli N, Butera NM, Younes N; GRADE Research Group. Optimization of Metformin in the GRADE Cohort: Effect on Glycemia and Body Weight. Diabetes Care. 2020 May;43(5):940-947. doi: 10.2337/dc19-1769. Epub 2020 Mar 5. PMID 32139384
- [Result] Wexler DJ, Krause-Steinrauf H, Crandall JP, Florez HJ, Hox SH, Kuhn A, Sood A, Underkofler C, Aroda VR; GRADE Research Group. Baseline Characteristics of Randomized Participants in the Glycemia Reduction Approaches in Diabetes: A Comparative Effectiveness Study (GRADE). Diabetes Care. 2019 Nov;42(11):2098-2107. doi: 10.2337/dc19-0901. Epub 2019 Aug 7. PMID 31391203
- [Result] Larkin ME, Nathan DM, Bebu I, Krause-Steinrauf H, Herman WH, Higgins JM, Tiktin M, Cohen RM, Lund C, Bergenstal RM, Johnson ML, Arends V; GRADE Research Group. Rationale and Design for a GRADE Substudy of Continuous Glucose Monitoring. Diabetes Technol Ther. 2019 Dec;21(12):682-690. doi: 10.1089/dia.2019.0202. Epub 2019 Sep 4. PMID 31393176
- [Result] Behringer-Massera S, Browne T, George G, Duran S, Cherrington A, McKee MD; GRADE Research Group. Facilitators and barriers to successful recruitment into a large comparative effectiveness trial: a qualitative study. J Comp Eff Res. 2019 Jul;8(10):815-826. doi: 10.2217/cer-2019-0010. Epub 2019 Aug 1. PMID 31368793
- [Result] Devchand R, Nicols C, Gallivan JM, Tiktin M, Krause-Steinrauf H, Larkin M, Tuncer DM; GRADE Research Group. Assessment of a National Diabetes Education Program diabetes management booklet: The GRADE experience. J Am Assoc Nurse Pract. 2017 May;29(5):255-263. doi: 10.1002/2327-6924.12445. Epub 2017 Feb 18. PMID 28213915
- [Result] Nathan DM, Buse JB, Kahn SE, Krause-Steinrauf H, Larkin ME, Staten M, Wexler D, Lachin JM; GRADE Study Research Group. Rationale and design of the glycemia reduction approaches in diabetes: a comparative effectiveness study (GRADE). Diabetes Care. 2013 Aug;36(8):2254-61. doi: 10.2337/dc13-0356. Epub 2013 May 20. PMID 23690531
- [Derived] Li JH, Szczerbinski L, Tripputi M, Liu H, Nam S, Mujica E, Emmanouilidou A, Wangden TY, Citko-Rojewska A, Konopka P, Czajkowski M, Huerta-Chagoya A, Vora M, Leong A, Meigs JB, Ng MY, Loos RJF, Pigeyre M, Gerstein HC, Moura FA, Lai YP, Bhatt DL, Marston NA, Ruff CT, Sabatine MS, Dawed AY, Pearson ER, Satin LS, den Hoed M, Kretowski A, Kahn SE, Younes N, Mercader JM, Florez JC. Common genetic variants near SLC2A2 and glycemic response to glimepiride in the GRADE comparative effectiveness clinical trial. medRxiv [Preprint]. 2025 Oct 8:2025.10.07.25336827. doi: 10.1101/2025.10.07.25336827. PMID 41282760
- [Derived] Natale P, Green SC, Tunnicliffe DJ, Pellegrino G, Toyama T, Strippoli GF. Glucagon-like peptide 1 (GLP-1) receptor agonists for people with chronic kidney disease and diabetes. Cochrane Database Syst Rev. 2025 Feb 18;2(2):CD015849. doi: 10.1002/14651858.CD015849.pub2. PMID 39963952
- [Derived] El-Damanawi R, Stanley IK, Staatz C, Pascoe EM, Craig JC, Johnson DW, Mallett AJ, Hawley CM, Milanzi E, Hiemstra TF, Viecelli AK. Metformin for preventing the progression of chronic kidney disease. Cochrane Database Syst Rev. 2024 Jun 4;6(6):CD013414. doi: 10.1002/14651858.CD013414.pub2. PMID 38837240

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: During a run-in period of 6 to 14 weeks before randomization, the metformin dose was increased to a minimum of 1000 mg per day, with a target maximal dose (one that could be taken without unacceptable side effects) of 2000 mg per day. Of the 7,850 participants consented for study run-in, 5,047 were randomized into the trial.
Groups:
- Glargine Insulin U-100: Glargine Insulin U-100 was administered daily at an initial dose of up to 20 U and adjusted according to glucose levels monitored by the participant and to avoid hypoglycemia.
- Glimepiride: Sulfonylurea glimepiride was increased from 1 to 2 mg to a maximum of 8 mg per day, administered in divided doses and adjusted according to glucose levels monitored by the participant and to avoid hypoglycemia.
- Liraglutide: GLP-1 analog liraglutide was initiated at a dose of 0.6 mg, with escalation to a maximum dose of 1.8 mg daily, depending on gastrointestinal side effects.
- Sitagliptin: DPP-4 inhibitor sitagliptin was initiated at a dose of 100 mg, with the dose adjusted according to kidney function.
Period: Overall Study
Arm/Group | Glargine Insulin U-100 | Glimepiride | Liraglutide | Sitagliptin
Started | 1263 | 1254 | 1262 | 1268
Completed | 1138 | 1142 | 1156 | 1144
Not Completed | 125 | 112 | 106 | 124

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Glargine Insulin U-100 | Glimepiride | Liraglutide | Sitagliptin | Total
Number analyzed (Participants) | 1263 | 1254 | 1262 | 1268 | 5047
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.0 (9.9) | 57.1 (10.1) | 57.4 (9.9) | 57.2 (10.1) | 57.2 (10.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 452 | 476 | 439 | 470 | 1837
  Male | 811 | 778 | 823 | 798 | 3210
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 33 | 30 | 40 | 34 | 137
  Asian | 34 | 47 | 47 | 54 | 182
  Native Hawaiian or Other Pacific Islander | 5 | 7 | 8 | 8 | 28
  Black or African American | 253 | 271 | 251 | 225 | 1000
  White | 837 | 808 | 815 | 854 | 3314
  More than one race | 82 | 71 | 82 | 84 | 319
  Unknown or Not Reported | 19 | 20 | 19 | 9 | 67
HbA1c [Mean (Standard Deviation); unit: %] | 7.5 (0.5) | 7.5 (0.5) | 7.5 (0.5) | 7.5 (0.5) | 7.5 (0.5)

OUTCOME MEASURES:

1. Primary Outcome: Time to HbA1c>=7%, While Receiving Metformin and the Randomly Assigned Glucose-lowering Study Medication
Description: The primary metabolic outcome is the time to primary failure defined as an HbA1c>=7% (53mmol/mol), subsequently confirmed, after addition of randomly assigned glucose-lowering medication at baseline.
Time Frame: Quarterly for 4 to 7 years
Measure: Median (Inter-Quartile Range); unit: years
Groups:
- Sitagliptin: DPP-4 inhibitor
Arm/Group | Glargine Insulin U-100 | Glimepiride | Liraglutide | Sitagliptin
Number analyzed (Participants) | 1263 | 1254 | 1262 | 1268
years | 1.3 [0.6 to 2.5] | 1.3 [0.6 to 2.3] | 1.5 [0.6 to 2.7] | 0.8 [0.5 to 2.0]

2. Secondary Outcome: Time to HbA1c>7.5%, While Receiving Metformin and the Randomly Assigned Glucose-lowering Study Medication.
Description: The secondary metabolic outcome is time to HbA1c>7.5% (58 mmol/mol), confirmed, after addition of randomly assigned glucose-lowering medication at baseline.
Time Frame: Quarterly, 4-6 years
Measure: Median (Inter-Quartile Range); unit: years
Groups:
- Glargine Insulin U-100: Insulin
- Glimepiride: Sulfonylurea
- Liraglutide: GLP-1 analog
Arm/Group | Glargine Insulin U-100 | Glimepiride | Liraglutide | Sitagliptin
Number analyzed (Participants) | 1263 | 1254 | 1262 | 1268
years | 2.1 [1.0 to 3.5] | 2.0 [1.1 to 3.3] | 2.2 [1.0 to 3.5] | 1.7 [0.8 to 3.0]

3. Primary Outcome: HbA1c>=7%, While Receiving Metformin and the Randomly Assigned Glucose-lowering Study Medication
Description: Number of participants who reached primary failure defined as an HbA1c>=7% (53mmol/mol), subsequently confirmed, after addition of randomly assigned glucose-lowering medication at baseline.
Time Frame: Quarterly, 4-7 years
Measure: Count of Participants; unit: Participants
Arm/Group | Glargine Insulin U-100 | Glimepiride | Liraglutide | Sitagliptin
Number analyzed (Participants) | 1263 | 1254 | 1262 | 1268
Participants | 852 | 908 | 860 | 981

4. Secondary Outcome: HbA1c>7.5%, While Receiving Metformin and the Randomly Assigned Glucose-lowering Study Medication.
Description: Number of participants who reached primary failure defined as an HbA1c>7.5% (58 mmol/mol), confirmed, after addition of randomly assigned glucose-lowering medication at baseline.
Time Frame: Quarterly for 4 to 7 years
Measure: Count of Participants; unit: Participants
Arm/Group | Glargine Insulin U-100 | Glimepiride | Liraglutide | Sitagliptin
Number analyzed (Participants) | 1263 | 1254 | 1262 | 1268
Participants | 498 | 633 | 583 | 697

ADVERSE EVENTS:
Time Frame: Quarterly for 4 to 7 years
Description: During the 6 to 14 weeks before randomization, a run-in period was used to determine eligibility into the study. Randomization occurred after successful completion of the run-in period. Adverse events prior to randomization were not considered part of the study and are not reported here.
Groups:
- Study Run-In (Metformin Only): During a run-in period of 6 to 14 weeks before randomization, the metformin dose was increased to a minimum of 1000 mg per day, with a target maximal dose (one that could be taken without unacceptable side effects) of 2000 mg per day.
Arm/Group | Glargine Insulin U-100 | Glimepiride | Liraglutide | Sitagliptin | Study Run-In (Metformin Only)
All-Cause Mortality (participants affected / at risk) | 42/1263 | 43/1254 | 27/1262 | 41/1268 | 0/7850
Serious Adverse Events (participants affected / at risk) | 259/1263 | 315/1254 | 204/1262 | 272/1268 | 1/7850
Other Adverse Events (participants affected / at risk) | 0/1263 | 0/1254 | 0/1262 | 0/1268 | 0/7850
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Glargine Insulin U-100 (N=1263) | Glimepiride (N=1254) | Liraglutide (N=1262) | Sitagliptin (N=1268) | Study Run-In (Metformin Only) (N=7850)
Severe Hypoglycemia (Metabolism and nutrition disorders) | 17 (21) | 28 (38) | 12 (13) | 9 (10) | 0 (0)
Heart failure (Cardiac disorders) | 26 (35) | 30 (49) | 14 (18) | 30 (56) | 0 (0)
Myocardial infarction (Cardiac disorders) | 30 (41) | 30 (33) | 21 (22) | 35 (37) | 0 (0)
Unstable angina (Cardiac disorders) | 9 (10) | 12 (14) | 7 (7) | 15 (17) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 10 (12) | 16 (18) | 11 (13) | 6 (6) | 0 (0)
Stent thrombosis (General disorders) | 0 (0) | 1 (1) | 2 (6) | 2 (2) | 0 (0)
Lactic Acidosis (Metabolism and nutrition disorders) | 6 (6) | 5 (5) | 6 (7) | 9 (11) | 0 (0)
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 (6) | 7 (7) | 3 (3) | 4 (4) | 0 (0)
Blood cancer other than leukemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 3 (3) | 2 (2) | 0 (0) | 0 (0)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 (5) | 5 (5) | 4 (4) | 5 (5) | 0 (0)
Cancer, Unknown primary (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
CNS/brain cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 5 (5) | 2 (2) | 4 (4) | 0 (0)
Esophageal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2) | 1 (1) | 1 (1) | 0 (0)
Gall Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Head/neck cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 4 (4) | 1 (1) | 3 (3) | 0 (0)
Kidney cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 5 (5) | 5 (5) | 9 (9) | 0 (0)
Leukemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 2 (2) | 2 (2) | 2 (2) | 0 (0)
Liver cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
Lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 7 (7) | 11 (11) | 7 (8) | 5 (5) | 0 (0)
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 3 (3) | 5 (5) | 5 (5) | 0 (0)
Other cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0) | 1 (1) | 3 (3) | 0 (0)
Other GI cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Ovarian cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pancreatic cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 (6) | 5 (5) | 3 (3) | 3 (3) | 1 (1)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 13 (13) | 22 (22) | 13 (13) | 14 (14) | 0 (0)
Skin (melanoma) cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 5 (6) | 6 (6) | 5 (5) | 0 (0)
Stomach cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2) | 2 (2) | 1 (1) | 0 (0)
Uterine cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (4) | 3 (3) | 4 (4) | 5 (5) | 0 (0)
Stroke (Nervous system disorders) | 23 (24) | 16 (18) | 19 (25) | 18 (22) | 0 (0)
Transient ischemic attack (Nervous system disorders) | 4 (4) | 8 (8) | 5 (6) | 5 (5) | 0 (0)
Coronary artery bypass graft (CABG) (Surgical and medical procedures) | 16 (16) | 20 (21) | 11 (11) | 25 (25) | 0 (0)
Interventional cardiology procedure (Surgical and medical procedures) | 40 (57) | 44 (58) | 23 (27) | 39 (46) | 0 (0)
Vascular/peripheral vascular intervention (Surgical and medical procedures) | 13 (14) | 14 (17) | 8 (16) | 7 (9) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (5):
  • Study Protocol (2017-03-17): https://cdn.clinicaltrials.gov/large-docs/43/NCT01794143/Prot_002.pdf
  • Statistical Analysis Plan: Manuscript - Microvascular and Cardiovascular Outcomes (OP2) (2022-04-08): https://cdn.clinicaltrials.gov/large-docs/43/NCT01794143/SAP_005.pdf
  • Statistical Analysis Plan: GRADE Study (2017-10-05): https://cdn.clinicaltrials.gov/large-docs/43/NCT01794143/SAP_001.pdf
  • Statistical Analysis Plan: Manuscript - Long Term Differences in Metabolic Status (OP1) (2022-03-22): https://cdn.clinicaltrials.gov/large-docs/43/NCT01794143/SAP_004.pdf
  • Informed Consent Form (2017-10-05): https://cdn.clinicaltrials.gov/large-docs/43/NCT01794143/ICF_003.pdf